CLINICAL TRIAL: NCT02965092
Title: Treatment of Relapsed or Refractory B-cell Malignancies by CD19 Chimeric Antigen Receptor (CAR)-Modified T Cells
Brief Title: CD19 Chimeric Antigen Receptor (CAR)-Modified T Cell Therapy in Treating Patients With B-cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan Sian Medical Technology Co., Ltd (Industry)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Jingzhou Central Hospital (Other); Xiangyang Central Hospital (Other); People Hospital Of Yichang (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-CD19-01
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Acute Lymphoblastic Leukemia; B Cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Second generation CAR-T cells (Experimental): Patients receive CD19 CAR-T cells transduced with a lentiviral vector on days 0, 1, and 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Genetic: Second generation CAR-T cells

INTERVENTIONS:
Genetic: Second generation CAR-T cells
  Other Names: CAR-T cells

SUMMARY:
This is a single arm, open-label, phase 1/2 study to evaluate the safety and efficacy of anti-CD19 CAR-T cells in patients with relapsed or refractory B cell Malignancies.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells (CAR-T cells) have the capabilities to recognize tumor associated antigen and kill tumor cells specifically. CAR-T therapy showed great effect on patients with relapsed or refractory B cell malignancies. CAR consists of single chain variable fragment (scFv) and activation domain of T cell. In preclinical study, the researchers constructed a second generation CAR containing CD137 costimulatory domain. This study aims to evaluate the safety and effectiveness of anti-CD19 CAR-T cells in patients with relapsed or refractory B cell Malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is pathologically and histologically confirmed as CD19 + B cell tumors, and has no effective treatment options currently, such as chemotherapy or autologous hematopoietic stem cell transplantation (auto-HSCT); or patients voluntarily choose CD19 CAR-T cells as a first treatment;
2. B cell hematological malignancies include the following three categories:

   * B-cell acute lymphocytic leukemia (B-ALL);
   * Indolent B-cell lymphoma (CLL, FL, MZL, LPL);
   * Aggressive B-cell lymphoma (DLBCL, BL, MCL);
3. < 70 years old;
4. Expected survival time > 6 months;
5. Female patients around childbearing age, negative pregnancy test before trial, and agreed to take effective contraceptive measures during the trial until the last visit;
6. Voluntarily participate in this experiment and sign informed consent by themself, or legally authorized representative.

Exclusion Criteria:

1. With a history of epilepsy or other central nervous system diseases;
2. Having graft-versus-host reaction, requires the use of immunosuppressants;
3. The presence of clinically significant cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within recent six months, or heart disease with cardiac function in any grade 3 (moderate) or 4 ( severe) (according to the New York Heart Association (NYHA) Functional Classification System);
4. Pregnant or lactating women (safety of this therapy for the unborn child is unknown);
5. Not curable active infection;
6. Patients with active hepatitis B or hepatitis C virus infection;
7. Combined use of systemic steroids within two weeks (except use of inhaled steroid recently or currently);
8. Using product of gene therapy before;
9. Creatinine> 2.5 mg / dl (221.0 umol/L); ALT / AST> 3 X the normal amount; Bilirubin> 2.0 mg / dl (34.2 umol/L);
10. Patients suffering from other uncontrolled diseases, and researchers believe that the patient is not suitable for trial;
11. Patients with HIV-infection;
12. Any situation that may increase the risk of patients or interfere with test results.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-12-02 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 5 years
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0)

SECONDARY OUTCOMES:
One-month remission rate | 1 month
  Response of B-ALL to CAR-T therapy was assessed on day 30 (±2), against the National Comprehensive Cancer Network (NCCN, Version 1.2015).
Overall survival | 5 years
  OS was calculated from the first CAR-T cell infusion to death or last follow-up (censored).
Event-free survival | 5 years
  EFS was calculated from the first CAR-T cell infusion to death, progression of the disease, relapse or gene recurrence, whichever came first, or last visit (censored).
Relapse-free survival | 5 years
  RFS was calculated from the first CAR-T cell infusion to relapse or last visit (censored).
Rate and quantity of anti-CD19 CAR-T cells in bone marrow cells and peripheral blood cells | 5 years
  In vivo (bone marrow and peripheral blood) rate and quantity of CAR-T cells were determined by means of flow cytometry and qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hu, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Du M, Mayombo RTM, Liu J, Zhang Y, Liao D, Hu Y, Mei H. The impact of obesity and its related underlying diseases on cytokine release syndrome and the efficacy of CAR-T therapy in treating B-cell malignancies. Ann Hematol. 2025 Mar;104(3):1887-1895. doi: 10.1007/s00277-025-06338-6. Epub 2025 Apr 8. PMID 40195173
- [Derived] Zhang Y, Zhou F, Wu Z, Li Y, Li C, Du M, Luo W, Kou H, Lu C, Mei H. Timing of Tocilizumab Administration Under the Guidance of IL-6 in CAR-T Therapy for R/R Acute Lymphoblastic Leukemia. Front Immunol. 2022 Jun 21;13:914959. doi: 10.3389/fimmu.2022.914959. eCollection 2022. PMID 35799791